CLINICAL TRIAL: NCT05031143
Title: Suprachoroidal Triamcinolone Acetonide Injection A Novel Therapy for Serous Retinal Detachment in Vogt-Koyanagi Harada's Disease
Brief Title: Suprachoroidal Triamcinolone Acetonide in Harada's Retinal Detachment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelshafy, Lecturer of Ophthalmology, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDASU-RECD-1234441
Record Dates: First submitted 2021-08-26; First posted 2021-09-01 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Vogt Koyanagi Harada Disease
Keywords: Vogt-koyanagi Harada, Suprachoroidal injection
MeSH Terms: conditions — Uveomeningoencephalitic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SCTA injection (n=6 eyes) (Active Comparator): Suprachoroidal Trimacinolone Acetonide injection 4mg/0.1ml, single dose, follow up for 6 months.
  Interventions: Drug: Suprachoroidal Triamcinolone acetonide injection for serous retinal detachment in VKH disease
- Non-injected eyes (Standard Treatment) (n=6 eyes) (No Intervention): Non-injected eyes on systemic steroids (standard treatment) and follow up for 6 months

INTERVENTIONS:
Drug: Suprachoroidal Triamcinolone acetonide injection for serous retinal detachment in VKH disease — Suprachoroidal steroid injection for management of serous retinal detachment in VKH disease
  Other Names: SCTA for Exudative RD in VKH disease
  Arms: SCTA injection (n=6 eyes)

SUMMARY:
Suprachoroidal injection, a novel technique for delivering ocular therapies, may facilitate targeted therapeutic delivery to the choroidal and retinal structures than intravitreal injection

DETAILED DESCRIPTION:
Suprachoroidal injection, a novel technique for delivering ocular therapies, may facilitate targeted therapeutic delivery to the choroidal and retinal structures than intravitreal injection. Yielding high levels of corticosteroid in the retinal and choroidal layers which was detectable for more than 3 months with limited exposure in the anterior segment. Triamcinolone acetonide is a synthetic corticosteroid formulated as an injectable suspension and has been evaluated in a number of trials to be 7.5 fold more potent anti-inflammatory than cortisone. Triamcinolone acetonide enhance tight junctions between endothelial cells thus reducing vessel leakage. It also has an angiostatic action by inhibition of vascular endothelial growth factor and has a useful effect on many inflammatory retinal diseases. The recommended dose of Triamcinolone acetonide injection is 4 mg/0.1 mL which was administrated in this study. The aim of this study was to assess the efficacy of suprachoroidal Triamcinolone acetonide injection (SCTA) as adjunctive therapy in the management of Vogt-Koyanagi Harada's (VKH) multiple serous retinal detachment (RD) and evaluate best corrected visual acuity (BCVA), intraocular pressure(IOP) and central foveal thickness (CFT) by Optical Coherence Tomography (OCT) in patients diagnosed as VKH at ophthalmology clinic, Benha University, EGYPT and Ebsar eye center, Benha, EGYPT.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed as VKH serous retinal detachment in the acute phase whom BCVA is not improving after 2 weeks from starting systemic steroids.

Exclusion Criteria:

* recent intraocular surgery.
* patients refuse to participate in the study.
* media opacity and other causes of serous retinal detachment than VKH.

Ages: 47 Years to 52 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity (LogMAR units) | 6 months after injection
  Changes in vision from baseline upto 6 months follow up

SECONDARY OUTCOMES:
Central Foveal Thickness measured by Optical Coherence Tomography | Upto 6 months after SCTA injection
  Changes in CFT during 6 months after injection

OTHER OUTCOMES:
Intraocular pressure measured by Goldmann applanation tonometry | 6 months after injection
  Changes in IOP during 6 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdelshafy, MD, Principal Investigator — Benha University, faculty of medicine; Marwa Abdelshafy, MD, Study Director — Benha University, faculty of medicine; Mohamed Anany, MD, Study Chair — Benha University, faculty of medicine
Locations (1):
- Ophthalmology department,Benha University and Ebsar eye center,Benha,EGYPT, Banhā, Qualiobeya, Egypt

IPD SHARING:
Plan to Share IPD: No